CLINICAL TRIAL: NCT00942448
Title: Efficacy and Safety Study of Diclofenac HPBCD 25, 50 mg/ml Administered as Single s.c. Dose, in the Treatment of Acute Moderate-to-severe Post-surgical Pain From Dental Surgery (Impacted 3rd Molar Extraction)
Brief Title: Evaluation of the Efficacy and Safety of Diclofenac HPBCD 25, 50 mg/ml in the Treatment of Post-surgical Pain Following Dental Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09PUK-DCsc04
Record Dates: First submitted 2009-07-17; First posted 2009-07-21 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2011-02

CONDITIONS: Dental Pain
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diclofenac HPBCD s.c. 25mg/ml (Experimental)
  Interventions: Drug: Diclofenac HPBCD
- Diclofenac HPBCD s.c. 50mg/ml (Experimental)
  Interventions: Drug: Diclofenac HPBCD
- Diclofenac HPBCD s.c. 75mg/ml (Active Comparator)
  Interventions: Drug: Diclofenac HPBCD
- Placebo s.c. (1ml) (Placebo Comparator)
  Interventions: Other: Placebo s.c.

INTERVENTIONS:
Drug: Diclofenac HPBCD — 1 single injection at day of dental surgical extraction
  Arms: Diclofenac HPBCD s.c. 25mg/ml
Drug: Diclofenac HPBCD — 1 single injection at day of dental surgical extraction
  Arms: Diclofenac HPBCD s.c. 50mg/ml
Drug: Diclofenac HPBCD — 1 single injection at day of dental surgical extraction
  Arms: Diclofenac HPBCD s.c. 75mg/ml
Other: Placebo s.c. — 1 single injection at day of dental surgical extraction
  Arms: Placebo s.c. (1ml)

SUMMARY:
The present study is proposed to evaluate the efficacy and safety of single doses of Diclofenac HPBCD subcutaneous (s.c.) (25 mg/1 ml and 50 mg/1 ml) in the treatment of acute moderate-to-severe pain after dental impaction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgical extraction of a single fully or partially impacted mandibular 3rd molar requiring bone removal.
* Patients experiencing moderate to severe post-operative pain within 6 hours from end of surgery.
* Pre-operative laboratory tests in the reference ranges or without clinically significant abnormalities as judged by the Investigator.

Exclusion Criteria:

* Surgery performed under general anaesthesia, or sedation.
* Complications occurring during the surgical procedure or in the period before randomisation as judged by the investigator.
* Acute local or systemic infection at the time of surgery that could confound the post-surgical evaluation.
* Patients with clinical signs of gastritis, gastro-duodenal ulcer, GI bleeding. Other GI disturbances or disease that in the opinion of the investigator could be negatively affected by the administration of NSAIDs.
* Clinical signs or history of coagulation disorders that could be negatively affected by NSAIDs administration.
* Hepatic or renal impairment.
* Patients with significant cardiac impairment, history of cerebrovascular disease, history or peripheral arterial disease, uncontrolled hypertension.
* Hypersensitivity to diclofenac or other NSAIDs or to one of the study medication components.
* Patients under chronic treatment with topical or systemic analgesics/NSAIDs.
* Patients under treatment with any medication that may affect the treatment efficacy evaluation.
* Patients under treatment with any medication whose concomitant use may be susceptible to interactions with diclofenac or may affect safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2009-09; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Dietrich, Prof, Principal Investigator — The school of dentistry, University of Birmingham
Locations (6):
- Poland (4):
  - Gabinet Stomatologiczny Bartek, Kobyłka
  - Centrum Leczenia Chorób Cywilizacyjnych, Warsaw
  - Niepubliczny Zakład Opieki Zdrowotnej, Warsaw
  - NZOZ Polimedica, Zgierz
- United Kingdom (2):
  - The School of Dentistry; University of Birmingham, Birmingham
  - Eastman Dental Institute, University College London, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients already scheduled for the surgical extraction of a single fully or partially impacted mandibular 3rd molar underwent a screening visit within 30 days from the scheduled date of surgery.
Pre-assignment Details: Patients under treatment with other analgesics, Major or minor tranquillizers, Muscle relaxant, Antihistamines, MAO inhibitors or corticosteroids had to undergo a wash out period prior to inclusion in the study.
Groups:
- Diclofenac HPBCD s.c. 25mg/ml; Diclofenac HPBCD s.c. 50mg/ml; Diclofenac HPBCD s.c. 75mg/ml: Diclofenac HPBCD : 1 single injection at day of dental surgical extraction
- Placebo s.c. (1ml): Placebo s.c. : 1 single injection at day of dental surgical extraction
Period: Overall Study
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. (1ml)
Started | 77 | 76 | 78 | 75
Completed | 77 | 76 | 78 | 75
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. (1ml) | Total
Number analyzed (Participants) | 77 | 76 | 78 | 75 | 306
Age Continuous [Mean (Standard Deviation); unit: years] | 30.7 (10.3) | 29.5 (8.68) | 30.2 (8.76) | 31.9 (11.3) | 30.56 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 48 | 46 | 44 | 184
  Male | 31 | 28 | 32 | 31 | 122

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Difference (PID) on a 0-100 VAS
Description: Pain intensity difference (PID) was derived by subtracting each pain intensity score (PI) from the baseline PI score (t0), where PI was assigned by the patient on a 0-100 mm VAS (from 0 = no pain to 100 = worst pain imaginable).
Time Frame: at 1.5 hours after treatment administration
Population: The reported number of analized participants were included in the ITT which was defined as all randomized patients who received the study medication and with at least one post-baseline efficacy evaluation within 1.5 hours post-dose (primary endpoint);
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. (1ml)
Number analyzed (Participants) | 77 | 76 | 78 | 75
mm | 36.5 [31.7 to 41.2] | 37.3 [32.6 to 42.1] | 37.7 [33.0 to 42.4] | 12.3 [7.44 to 17.1]
Statistical Analysis 1: Comparison: Diclofenac HPBCD s.c. 25mg/ml vs Placebo s.c. (1ml); The sample size calculation was based on a hypothesis of superiority of diclofenac HPBCD s.c. 25mg/ml and 50 mg/ml compared to Placebo with regard to the primary efficacy variable (PID at 1.5 hours following drug administration). A sample size of 60 in each group had 95% power to detect a difference between diclofenac HPBCD s.c. 25 mg/ml and placebo in means of 15 mm, assuming that the common standard deviation was 22.5 and using a two group t-test with a 0.05 two-sided significance level; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 24.2
Statistical Analysis 2: Comparison: Diclofenac HPBCD s.c. 50mg/ml vs Placebo s.c. (1ml); Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Final Values) = 25.1, 95% CI 2-sided [18.4 to 31.7]

2. Secondary Outcome: PID
Description: as for outcome 1
Time Frame: at 15 minutes post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. 1ml
Number analyzed (Participants) | 77 | 76 | 78 | 75
mm | 8.39 (14.1) | 8.28 (13.7) | 9.46 (15.7) | 1.59 (11.3)

3. Secondary Outcome: PID
Description: as for outcome 1
Time Frame: at 30 minutes post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. 1ml
Number analyzed (Participants) | 77 | 76 | 78 | 75
mm | 15.9 (16.4) | 18.5 (19.5) | 18.6 (18.9) | 4.68 (17.2)

4. Secondary Outcome: PID
Description: as for outcome 1
Time Frame: at 45 minutes post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. 1ml
Number analyzed (Participants) | 77 | 76 | 78 | 75
mm | 24.7 (17.9) | 27.5 (22.1) | 27.8 (19.0) | 9.00 (20.9)

5. Secondary Outcome: PID
Description: as for outcome 1
Time Frame: at 60 minutes post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. 1ml
Number analyzed (Participants) | 77 | 76 | 78 | 75
mm | 30.7 (18.0) | 34.6 (23.0) | 34.6 (18.7) | 15.3 (24.0)

6. Secondary Outcome: PID
Description: as for outcome 1
Time Frame: at 90 minutes post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. 1ml
Number analyzed (Participants) | 77 | 76 | 78 | 75
mm | 36.2 (19.2) | 40.1 (20.8) | 39.0 (18.9) | 18.0 (26.0)

7. Secondary Outcome: PID
Description: as for outcome 1
Time Frame: at 2 hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. 1ml
Number analyzed (Participants) | 77 | 76 | 78 | 75
mm | 38.8 (19.1) | 43.9 (20.4) | 42.5 (18.2) | 26.5 (25.1)

8. Secondary Outcome: PID
Description: as for outcome 1
Time Frame: at 3 hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. 1ml
Number analyzed (Participants) | 77 | 76 | 78 | 75
mm | 41.2 (20.0) | 45.5 (21.0) | 45.6 (19.2) | 25.3 (26.8)

9. Secondary Outcome: PID
Description: as for outcome 1
Time Frame: at 4 hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. 1ml
Number analyzed (Participants) | 77 | 76 | 78 | 75
mm | 38.1 (21.2) | 46.3 (21.8) | 48.0 (18.6) | 29.1 (26.8)

10. Secondary Outcome: PID
Description: as for outcome 1
Time Frame: at 5 hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. 1ml
Number analyzed (Participants) | 77 | 76 | 78 | 75
mm | 37.5 (20.9) | 42.2 (23.8) | 45.6 (18.3) | 31.8 (22.0)

11. Secondary Outcome: PID
Description: as for outcome 1
Time Frame: at 6 hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. 1ml
Number analyzed (Participants) | 77 | 76 | 78 | 75
mm | 41.5 (19.8) | 40.9 (23.4) | 41.7 (22.4) | 36.5 (14.6)

12. Secondary Outcome: PID
Description: as for outcome 1
Time Frame: at 7 hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. 1ml
Number analyzed (Participants) | 77 | 76 | 78 | 75
mm | 43.2 (17.9) | 41.6 (24.3) | 43.0 (19.2) | 39.1 (13.5)

13. Secondary Outcome: PID
Description: as for outcome 1
Time Frame: at 8 hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. 1ml
Number analyzed (Participants) | 77 | 76 | 78 | 75
mm | 45.0 (15.7) | 43.8 (25.2) | 43.6 (17.5) | 37.0 (14.3)

14. Primary Outcome: Pain Intensity Difference (PID) on a 0-100 VAS
Description: as for outcome 1
Time Frame: at 1.5 hours after treatment administration
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. (1ml)
Number analyzed (Participants) | 77 | 76 | 78 | 75
mm | 36.5 [31.7 to 41.2] | 37.3 [32.6 to 42.1] | 37.7 [33.0 to 42.4] | 12.3 [7.44 to 17.1]
Statistical Analysis 1: Comparison: Diclofenac HPBCD s.c. 25mg/ml vs Placebo s.c. (1ml); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 24.2, 95% CI 2-sided [17.6 to 30.8]
Statistical Analysis 2: Comparison: Diclofenac HPBCD s.c. 50mg/ml vs Placebo s.c. (1ml); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 25.1, 95% CI 2-sided [18.4 to 31.7]

ADVERSE EVENTS:
Arm/Group | Diclofenac HPBCD s.c. 25mg/ml | Diclofenac HPBCD s.c. 50mg/ml | Diclofenac HPBCD s.c. 75mg/ml | Placebo s.c. (1ml)
Serious Adverse Events (participants affected / at risk) | 0/77 | 1/76 | 0/78 | 0/75
Other Adverse Events (participants affected / at risk) | 3/77 | 3/76 | 5/78 | 5/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac HPBCD s.c. 25mg/ml (N=77) | Diclofenac HPBCD s.c. 50mg/ml (N=76) | Diclofenac HPBCD s.c. 75mg/ml (N=78) | Placebo s.c. (1ml) (N=75)
gingival abscess (Infections and infestations) | 0 (0) | 1 (76) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac HPBCD s.c. 25mg/ml (N=77) | Diclofenac HPBCD s.c. 50mg/ml (N=76) | Diclofenac HPBCD s.c. 75mg/ml (N=78) | Placebo s.c. (1ml) (N=75)
Headache (Nervous system disorders) | 3 (5) | 3 (3) | 5 (6) | 5 (6)

LIMITATIONS AND CAVEATS:
No limitations of the trial have been detected

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less